CLINICAL TRIAL: NCT00383656
Title: Pulsatile GnRH in Anovulatory Infertility
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Janet E. Hall, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1999-P-004396; 5U54HD028138 (NIH)
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Hypogonadotropic Hypogonadism; Amenorrhea; Kallmann's Syndrome
Keywords: gonadotropin releasing hormone; GnRH deficiency; hypothalamic amenorrhea; hypogonadotropic hypogonadism; Kallman's syndrome; infertility
MeSH Terms: conditions — Hypogonadism; Amenorrhea; Kallmann Syndrome; Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pulsatile GnRH (Experimental): All participants will be administered GnRH intravenously by means of a portable infusion pump that delivers boluses at specific intervals.
  Interventions: Drug: GnRH; Device: Pump

INTERVENTIONS:
Drug: GnRH — 75 ng/kg GnRH IV
  Other Names: gonaodtropin releasing hormone; GnRH pump
Device: Pump — portable, infusion pump for GnRH
  Other Names: mini-infusion pump

SUMMARY:
The purpose of this study is to explore the effects of synthetic gonadotropin-releasing hormone (GnRH) upon the pituitary and ovaries of women with infertility. Women diagnosed with GnRH deficiency, hypothalamic amenorrhea or acquired hypogonadic hypogonadism, will participate in this study. It is hoped that administration of GnRH will lead to proper stimulation of the pituitary gland and to normal ovulation and menstruation.

**WE ARE CURRENTLY RECRUITING ONLY WOMEN WITH A DIAGNOSIS OF IDIOPATHIC HYPOGONADIC HYPOGONADISM (IHH)**

Pulsatile GnRH has been approved by the FDA for use in women with primary amenorrhea due to complete GnRH deficiency. The overall goals of this protocol are to continue to use pulsatile GnRH in GnRH-deficient and other anovulatory women for ovulation induction and to examine specific physiologic hypotheses, which can only be addressed in this patient population.

DETAILED DESCRIPTION:
In comparison to the use of exogenous gonadotropins, pulsatile administration of GnRH has many theoretical advantages for ovulation induction, including; 1) the ability to use the patients' own gonadotropins for ovarian stimulation; 2) the ability to treat anovulatory defects at their appropriate level, which most commonly is hypothalamic; 3) the ability to maintain normal ovarian-pituitary feedback mechanisms to restrain endogenous FSH secretion, as occurs normally in species that ovulate a single egg per cycle; 4) a resultant decrease in the risks of multiple gestations and hyperstimulation; and 5) a decreased need for intensive monitoring of ovarian function with an attendant decrease in costs.

When synthetic GnRH first became available for clinical study, there was not yet an adequate understanding of the physiology of GnRH secretion in the human to support its potential therapeutic application. As a result, early attempts at ovulation induction were unsuccessful. It was soon appreciated that an episodic mode of delivery was essential for normal pituitary stimulation by GnRH. Studies by our group and others which defined the frequency of pulsatile GnRH secretion in normal women at different stages of the menstrual were then key to designing a physiologic program of pulsatile GnRH administration that resulted in successful ovulation induction in patients with GnRH deficiency. Additional studies demonstrated that which replacement of GnRH using the subcutaneous route was adequate to reproduce normal physiology in GnRH-deficient men, the intravenous route was superior in women. We have now determined the dose of GnRH which is appropriate for the majority of women as 75 ng/kg, a dose which induces ovulation of a single dominant follicle, followed by normal luteal phase dynamics.

A number of investigators including us have sought to define the specific subgroups likely to achieve the greatest benefit from this form of therapy. However, there are many questions which remain unanswered and that we are currently addressing. We are specifically interested in understanding why there is variability in the dose of GnRH required by apparently GnRH-deficient women.

It is important to note that minors have been included in this protocol, as many patients are extremely anxious to know whether they respond normally to pulsatile GnRH even though they may not be interested in conceiving at the time. This is particularly true of patients who have survived childhood cancers and associated surgery and/or radiation in whom a normal response to pulsatile GnRH can be a very positive experience.

ELIGIBILITY:
Inclusion Criteria:

* Women and minors with GnRH deficiency or idiopathic hypogonadotropic hypogonadism (IHH) will have a history of primary amenorrhea, no evidence of abnormalities in other hormonal axes, a deficient pattern of luteinizing hormone (LH) and/or free alpha subunit (FAS) secretion on baseline sampling and a normal cranial CT or MRI.
* Women and minors with hypothalamic amenorrhea will have a history of secondary amenorrhea of at least six months duration with low or normal gonadotropins or a history of primary amenorrhea in the presence of pulsatile patterns of LH or FAS on baseline frequent sampling studies, BMI > 18 kg/m2 and normal testosterone and prolactin levels.
* Women and minors with acquired hypogonadotropic hypogonadism will have a history of hypothalamic or pituitary tumor treated with surgery alone or in combination with radiotherapy or a history of hypothalamic irradiation as adjunctive therapy for leukemia or craniofacial neoplasms. There must be a minimum of 2 years since irradiation and no gonadal radiation. For the previous two months, patients will be euthyroid on thyroid replacement if needed, normoprolactinemic on dopamine agonists if needed, and receiving physiologic glucocorticoid replacement if needed.

Subjects will be otherwise healthy women and female minors between the ages of 16 and 45 years who have not been on gonadal steroid preparations for at least 1 month. Subjects will have normal complete blood count (hemoglobin greater than or equal to 11.5gm/dl) and thyroid function tests and a negative pregnancy test.

Exclusion Criteria:

Mitral valve prolapse with ballooning of the mitral valve will be cause for exclusion of the patient from intravenous GnRH treatment.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Estimated)
Dates: Start 1989-01; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
ovulation | 1 pulsatile GnRH cycle
  LH surge or luteal phase progesterone > 5 ng/dL

SECONDARY OUTCOMES:
pregnancy | 6 weeks
  serum HCG indicative of pregnancy

OTHER OUTCOMES:
LH | 1st 7 days of treatment
  LH levels from days 1-7of treatment of treatment
FSH | 1st 7 days of treatment
  FSH levels from days 1-7 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Hall, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared across MGH and NIH protocols to which the participant consents.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: For the duration of the study.
Access Criteria: must be approved by the study PI

REFERENCES:
- [Background] Martin K, Santoro N, Hall J, Filicori M, Wierman M, Crowley WF Jr. Clinical review 15: Management of ovulatory disorders with pulsatile gonadotropin-releasing hormone. J Clin Endocrinol Metab. 1990 Nov;71(5):1081A-1081G. doi: 10.1210/jcem-71-5-1081. PMID 2229271
- [Background] Martin KA, Hall JE, Adams JM, Crowley WF Jr. Comparison of exogenous gonadotropins and pulsatile gonadotropin-releasing hormone for induction of ovulation in hypogonadotropic amenorrhea. J Clin Endocrinol Metab. 1993 Jul;77(1):125-9. doi: 10.1210/jcem.77.1.8325934.
- [Background] Santoro N, Wierman ME, Filicori M, Waldstreicher J, Crowley WF Jr. Intravenous administration of pulsatile gonadotropin-releasing hormone in hypothalamic amenorrhea: effects of dosage. J Clin Endocrinol Metab. 1986 Jan;62(1):109-16. doi: 10.1210/jcem-62-1-109. PMID 3079597
- [Background] Homburg R, Eshel A, Armar NA, Tucker M, Mason PW, Adams J, Kilborn J, Sutherland IA, Jacobs HS. One hundred pregnancies after treatment with pulsatile luteinising hormone releasing hormone to induce ovulation. BMJ. 1989 Mar 25;298(6676):809-12. doi: 10.1136/bmj.298.6676.809. PMID 2496866
- [Background] Filicori M, Flamigni C, Meriggiola MC, Ferrari P, Michelacci L, Campaniello E, Valdiserri A, Cognigni G. Endocrine response determines the clinical outcome of pulsatile gonadotropin-releasing hormone ovulation induction in different ovulatory disorders. J Clin Endocrinol Metab. 1991 May;72(5):965-72. doi: 10.1210/jcem-72-5-965. PMID 1902487
- [Background] Filicori M, Flamigni C, Meriggiola MC, Cognigni G, Valdiserri A, Ferrari P, Campaniello E. Ovulation induction with pulsatile gonadotropin-releasing hormone: technical modalities and clinical perspectives. Fertil Steril. 1991 Jul;56(1):1-13. doi: 10.1016/s0015-0282(16)54407-0. No abstract available. PMID 2065788
- [Background] Hall JE, Martin KA, Whitney HA, Landy H, Crowley WF Jr. Potential for fertility with replacement of hypothalamic gonadotropin-releasing hormone in long term female survivors of cranial tumors. J Clin Endocrinol Metab. 1994 Oct;79(4):1166-72. doi: 10.1210/jcem.79.4.7962290.
- [Background] Seminara SB, Beranova M, Oliveira LM, Martin KA, Crowley WF Jr, Hall JE. Successful use of pulsatile gonadotropin-releasing hormone (GnRH) for ovulation induction and pregnancy in a patient with GnRH receptor mutations. J Clin Endocrinol Metab. 2000 Feb;85(2):556-62. doi: 10.1210/jcem.85.2.6357. PMID 10690855
- [Background] Lavoie HB, Martin KA, Taylor E, Crowley WF, Hall JE. Exaggerated free alpha-subunit levels during pulsatile gonadotropin-releasing hormone replacement in women with idiopathic hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 1998 Jan;83(1):241-7. doi: 10.1210/jcem.83.1.4488. PMID 9435449
- [Background] Nestler JE, Jakubowicz DJ, Evans WS, Pasquali R. Effects of metformin on spontaneous and clomiphene-induced ovulation in the polycystic ovary syndrome. N Engl J Med. 1998 Jun 25;338(26):1876-80. doi: 10.1056/NEJM199806253382603. PMID 9637806
- [Background] De Leo V, la Marca A, Ditto A, Morgante G, Cianci A. Effects of metformin on gonadotropin-induced ovulation in women with polycystic ovary syndrome. Fertil Steril. 1999 Aug;72(2):282-5. doi: 10.1016/s0015-0282(99)00208-3. PMID 10438996
- [Background] Hopkins CC, Hall JE, Santoro NF, Martin KA, Filicori M, Crowley WF Jr. Closed intravenous administration of gonadotropin-releasing hormone: safety of extended peripheral intravenous catheterization. Obstet Gynecol. 1989 Aug;74(2):267-70. PMID 2664612
- [Background] Coetzee EJ, Jackson WP. Pregnancy in established non-insulin-dependent diabetics. A five-and-a-half year study at Groote Schuur Hospital. S Afr Med J. 1980 Nov 15;58(20):795-802. PMID 6777880
- [Background] Coetzee EJ, Jackson WP. Oral hypoglycaemics in the first trimester and fetal outcome. S Afr Med J. 1984 Apr 21;65(16):635-7. PMID 6369573
- [Derived] Delaney A, Volochayev R, Meader B, Lee J, Almpani K, Noukelak GY, Henkind J, Chalmers L, Law JR, Williamson KA, Jacobsen CM, Buitrago TP, Perez O, Cho CH, Kaindl A, Rauch A, Steindl K, Garcia JE, Russell BE, Prasad R, Mondal UK, Reigstad HM, Clements S, Kim S, Inoue K, Arora G, Salnikov KB, DiOrio NP, Prada R, Capri Y, Morioka K, Mizota M, Zechi-Ceide RM, Kokitsu-Nakata NM, Tonello C, Vendramini-Pittoli S, da Silva Dalben G, Balasubramanian R, Dwyer AA, Seminara SB, Crowley WF, Plummer L, Hall JE, Graham JM, Lin AE, Shaw ND. Insight Into the Ontogeny of GnRH Neurons From Patients Born Without a Nose. J Clin Endocrinol Metab. 2020 May 1;105(5):1538-51. doi: 10.1210/clinem/dgaa065. PMID 32034419
- [Derived] Abel BS, Shaw ND, Brown JM, Adams JM, Alati T, Martin KA, Pitteloud N, Seminara SB, Plummer L, Pignatelli D, Crowley WF Jr, Welt CK, Hall JE. Responsiveness to a physiological regimen of GnRH therapy and relation to genotype in women with isolated hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 2013 Feb;98(2):E206-16. doi: 10.1210/jc.2012-3294. Epub 2013 Jan 22. PMID 23341491
- See also: MGH Reproductive Endocrine Unit — http://www.mgh.harvard.edu/reproendo/pages/reu_currentresearch.htm